CLINICAL TRIAL: NCT00532103
Title: Suicide Assessment Methodology Study (SAMS)
Brief Title: Assessing Treatment Emergent Suicidal Ideation in Patients With Major Depression
Acronym: SAMS
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Madhukar H. Trivedi, M.D., The University of Texas Southwestern Medical Center
Other Study IDs: N01 MH90003-01; DSIR AT; N01MH90003 (NIH)
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Depression
Keywords: Suicidal Ideation; Major Depressive Disorder; Suicide Risk; Antidepressant Medication
MeSH Terms: conditions — Depression; Suicidal Ideation; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will develop a new methodology to evaluate any treatment-emergent suicidal ideation that might occur when an antidepressant treatment has been started and/or during times when doses are increased in patients with major depressive disorder.

DETAILED DESCRIPTION:
This is a pilot study to begin to develop a measurement procedure to help guide the clinical management of suicide risk in people beginning a type of antidepressant medication called a selective serotonin reuptake inhibitor (SSRI). The goals of the study are: 1) to identify the best method and assessment measures to evaluate the severity of suicidal ideation, 2) to determine the appropriate frequency and duration of assessment required to adequately evaluate this suicidal ideation, 3) to evaluate the presence of symptoms that are associated with suicidal ideation (such as anxiety, panic attacks, difficulty in sleeping) and 4) to identify the most critical time periods during which suicidal ideation appears or worsens (such as how long after initiation of treatment or dosage increase).

In all, 300 adult participants with major depressive disorder (MDD), between the ages of 18 and 75, may be enrolled at primary and psychiatric care sites across the US. All patients will be treated with an SSRI for eight weeks. The choice of SSRI used in treatment will be chosen by the study physician at each site. For this study, physicians will choose from the following six SSRIs: citalopram, escitalopram, sertraline, paroxetine, paroxetine-CR, and fluoxetine.

Patients beginning an SSRI for MDD in "real world" psychiatric and primary care settings, will have clinic visits and receive evaluations of their symptoms of depression, side effects, suicidal thinking and symptoms that are thought to be associated with suicidal risk, every other week for eight weeks. They will be evaluated by phone for symptoms and side effects each week they do not come to the clinic. They will also receive phone calls three times a week for the first two weeks of the study, after beginning the antidepressant, and after a dose increase to evaluate suicide risk.

ELIGIBILITY:
Inclusion Criteria:

ONLY PATIENTS BEING TREATED AT THE PARTICIPATING CLINICS ARE ELIGIBLE FOR THIS STUDY

* Patients must be enrolled at the primary or specialty care site, and be planning to continue living in the area of that clinic throughout the study
* Patients must be 18-75 years old
* Patients must meet clinical criteria for MDD, based on clinical interview and DSM IV MDD checklist
* Screening HAM-D17 score greater than or equal to 14
* Patients must give written informed consent
* Patients with and without current suicidal ideation may be included in the study
* Patients must not have taken antidepressant medication for at least 2 weeks prior to screen (or 4 weeks in the case of fluoxetine).

Exclusion Criteria:

* Current substance abuse or dependence
* Two past SSRI treatment failures within the current episode, or last 2 years if chronic.
* Patients with a current Axis I diagnosis of Bipolar disorder or Schizophrenia
* Patients with a current Primary Axis I diagnosis of Obsessive-Compulsive disorder, Anorexia Nervosa or Bulimia.
* Women who are sexually active and who are not using adequate contraception, or who are pregnant, trying to become pregnant, or breast feeding.
* Patients with general medical conditions that contraindicate antidepressant medications
* Patients whose clinical status requires inpatient treatment at the time of baseline interview.
* Patients who cannot read and understand English since all research instruments are not yet translated and validated in Spanish or other languages.
* Some reports of SSRI-induced akathisia-like states have found them to be more highly correlated with either concurrent or previous treatment with a neuroleptic, even in patients with no history of movement disorders therefore, patients who have taken an anti-psychotic medication within 4 months of the screening visit will be excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifteen primary care and specialty care clinics across the country.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center; Stephen R. Wisniewski, PhD, Study Director — University of Pittsburgh; Diane Warden, PhD, MBA, Study Director — University of Texas Southwestern Medical Center; Kathy Shores-Wilson, PhD, Study Director — University of Texas Southwestern Medical Center; David W. Morris, PhD, Study Director — University of Texas Southwestern Medical Center
Locations (15):
- United States (15):
  - Tuscalossa VA Mental Health Clinic, Tuscaloosa, Alabama
  - Harbor UCLA Family Health Care Center, Harbor City, California
  - UCLA Internal Medicine Clinic, Los Angeles, California
  - Veterans Affairs Medical Center/FIRM Primary Care Clinic, San Diego, California
  - Northwestern Psychiatric Outpatient Treatment Care Center, Chicago, Illinois
  - Clinical Research Institute, Wichita, Kansas
  - MGH/Northshore Medical Center (Salem Psychiatric Facility), Salem, Massachusetts
  - General Psychiatric Ambulatory Clinic, Ann Arbor, Michigan
  - Irving Goldman Primary Care at North Shore Hospital, New York, New York
  - UNC Chapel Hill Adult Diagnostic & Treatment Clinic, Chapel Hill, North Carolina
  - Laureate Psychiatric Clinic and Hospital, Tulsa, Oklahoma
  - Bellefield Clinic of WPIC, Pittsburgh, Pennsylvania
  - Vine Hill Community Clinic, Nashville, Tennessee
  - UT Southwestern Family Medicine Clinic, Dallas, Texas
  - VCU Outpatient Psychiatry Clinic, Richmond, Virginia

REFERENCES:
- [Derived] Jha MK, Minhajuddin A, South C, Rush AJ, Trivedi MH. Irritability and Its Clinical Utility in Major Depressive Disorder: Prediction of Individual-Level Acute-Phase Outcomes Using Early Changes in Irritability and Depression Severity. Am J Psychiatry. 2019 May 1;176(5):358-366. doi: 10.1176/appi.ajp.2018.18030355. Epub 2019 Mar 29. PMID 30922100
- [Derived] Gollan JK, Fava M, Kurian B, Wisniewski SR, Rush AJ, Daly E, Miyahara S, Trivedi MH. What are the clinical implications of new onset or worsening anxiety during the first two weeks of SSRI treatment for depression? Depress Anxiety. 2012 Feb;29(2):94-101. doi: 10.1002/da.20917. Epub 2011 Dec 6. PMID 22147631
- [Derived] Trivedi MH, Wisniewski SR, Morris DW, Fava M, Kurian BT, Gollan JK, Nierenberg AA, Warden D, Gaynes BN, Luther JF, Rush AJ. Concise Associated Symptoms Tracking scale: a brief self-report and clinician rating of symptoms associated with suicidality. J Clin Psychiatry. 2011 Jun;72(6):765-74. doi: 10.4088/JCP.11m06840. PMID 21733477
- [Derived] Trivedi MH, Wisniewski SR, Morris DW, Fava M, Gollan JK, Warden D, Nierenberg AA, Gaynes BN, Husain MM, Luther JF, Zisook S, Rush AJ. Concise Health Risk Tracking scale: a brief self-report and clinician rating of suicidal risk. J Clin Psychiatry. 2011 Jun;72(6):757-64. doi: 10.4088/JCP.11m06837. PMID 21733476
- [Derived] Warden D, Trivedi MH, Wisniewski SR, Kurian B, Zisook S, Kornstein SG, Friedman ES, Miyahara S, Leuchter AF, Fava M, Rush AJ. Early adverse events and attrition in selective serotonin reuptake inhibitor treatment: a suicide assessment methodology study report. J Clin Psychopharmacol. 2010 Jun;30(3):259-66. doi: 10.1097/JCP.0b013e3181dbfd04. PMID 20473060